CLINICAL TRIAL: NCT07067294
Title: Effect of Low-Level Light Therapy on Ocular Surface Parameters in Patients Undergoing Cataract Surgery: A Randomized Controlled Clinical Trial
Brief Title: Effect of Low-Level Light Therapy on Ocular Surface Parameters in Patients Undergoing Cataract Surgery
Acronym: LLLT-Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Timofte Zorila Mihaela Madalina, Dr, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Grigore T. Popa n.54/290724
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye; Meibomian Gland Dysfunction (Disorder); Ocular Surface Disease
Keywords: Dry eye disease; LLLT; Photobiomodulation
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, single-masked, parallel-group trial. Eligible participants undergoing cataract surgery are randomly assigned in a 1:1 ratio to receive either low-level light therapy (LLLT) or a sham treatment. Interventions are administered perioperatively (1 week before and 1 week after surgery), and all clinical outcomes are assessed at baseline, 1 week, 1 month and 6 months postoperatively. Participants remain in their assigned group for the duration of the study, with no crossover between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLLT Group (Experimental): A total of 50 patients were randomized to the low-level light therapy (LLLT) group. All participants underwent standard cataract surgery and received two sessions of periocular LLLT using the Eye-light® device (Espansione Group, Italy): one session one week before surgery and another one week after. The treatment was delivered through a wearable mask emitting polychromatic red and near-infrared light, targeting the eyelids and meibomian glands.
  Of the 50 randomized patients, 3 were lost to follow-up and 2 discontinued the intervention due to postoperative complications. Ultimately, 45 patients completed the full study protocol and were included in the final analysis. Ocular surface assessments were performed at baseline, 1 week, 1 month, and 6 months postoperatively to evaluate the effects of LLLT on tear film quality, inflammation, and meibomian gland function.
  Interventions: Device: Low-Level Light Therapy
- Sham Group (Sham Comparator): A total of 48 patients were randomized to the sham group. These participants underwent standard cataract surgery and received two perioperative sessions of a simulated light-based treatment, one administered one week before and one week after surgery. The procedure mimicked the experience of the active LLLT intervention, using the same mask device without activation of the therapeutic light emission.
  Of the 48 enrolled participants, 2 were lost to follow-up and 2 discontinued due to postoperative complications. A total of 44 patients completed the full protocol and were included in the final analysis. Clinical assessments were conducted at the same time points as the active treatment group-baseline, 1 week, 1 month, and 6 months postoperatively-to evaluate tear film function, ocular surface condition, and meibomian gland performance.
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: Low-Level Light Therapy — The intervention consists of non-invasive periocular photobiomodulation using the Eye-light® device (Espansione Group, Italy), which delivers low-level polychromatic red and near-infrared light (600-1200 nm) through a specially designed mask. Participants receive two 15-minute sessions, one 7 days before and one 7 days after cataract surgery.
  The treatment is designed to stimulate meibomian gland activity, improve tear film stability, reduce ocular surface inflammation.
  This protocol is unique compared to standard treatments for dry eye because it targets cellular mitochondrial activity to enhance tissue repair and anti-inflammatory effects. It is non-pharmacological, non-contact, and well-tolerated, making it suitable for perioperative application. The light is delivered through closed eyelids, ensuring safety and comfort, and the device used is CE-marked for ophthalmic applications.
  Arms: LLLT Group
Device: Sham (No Treatment) — Sham-treated controls underwent the same procedural setup as the active treatment group, using the Eye-light® device (Espansione Group, Italy). However, instead of delivering therapeutic levels of light energy, the device operated in demo light mode, emitting less than 30% of the full treatment power. This setting simulated the visual and sensory experience of a low-level light therapy (LLLT) session without delivering biologically effective photobiomodulation.
  The sham intervention included two 15-minute sessions: one administered 7 days before cataract surgery and one 7 days after. This approach allowed for masking of participants and investigators to minimize bias, while ensuring that patients in the control group received no active therapeutic exposure.
  Arms: Sham Group

SUMMARY:
This randomized, controlled clinical trial investigates the perioperative use of low-level light therapy (LLLT) to prevent or reduce signs and symptoms of dry eye disease (DED) in patients undergoing cataract surgery. DED is a prevalent postoperative complication associated with ocular surface inflammation, meibomian gland dysfunction, and tear film instability, which can compromise visual outcomes and patient satisfaction.

The study enrolled adult patients scheduled for phacoemulsification, with baseline evidence of mild-to-moderate ocular surface disease. Participants were randomly assigned to receive either LLLT via a polychromatic light-emitting mask (Eye-light® ) or a sham device, administered one week before and one week after surgery. The LLLT protocol is designed to photobiomodulate eyelid and periocular tissues to enhance meibomian gland function and reduce subclinical inflammation.

Clinical assessments were conducted at baseline, one week, and six months postoperatively. The primary endpoint was the change in Ocular Surface Disease Index (OSDI) score at one and six months. Secondary endpoints included tear film stability (TBUT), Schirmer I test, corneal staining, tear osmolarity, and tear inflammatory and reparative biomarkers. The study also evaluated the safety and tolerability of the LLLT intervention.

This is the first prospective study assessing the role of perioperative LLLT in mitigating post-cataract ocular surface disease in consecutive patients. The findings may support the integration of LLLT in perioperative ocular surface management protocols.

DETAILED DESCRIPTION:
This single-center, randomized, single-masked, parallel-group clinical trial was conducted to evaluate the efficacy and safety of low-level light therapy (LLLT) in the perioperative management of dry eye disease (DED) in patients undergoing cataract surgery. The study was carried out at the Department of Ophthalmology, University of Medicine and Pharmacy "Grigore T. Popa" (Iași, Romania) in accordance with the Declaration of Helsinki and ICH-GCP guidelines.

Dry eye disease is a multifactorial disorder characterized by tear film instability and ocular surface inflammation. Cataract surgery is known to transiently exacerbate or precipitate DED through mechanisms including disruption of corneal nerves, exposure to surgical light and irrigation, and postoperative medication use. This can impair visual rehabilitation and reduce patient satisfaction with surgical outcomes, particularly in individuals with pre-existing ocular surface dysfunction.

LLLT is a non-invasive photobiomodulation technique that delivers low-intensity, polychromatic red and near-infrared light to target mitochondrial cytochromes and promote cellular activity. Its application in ophthalmology has shown potential to improve meibomian gland function, enhance tear film stability, and downregulate inflammatory cytokines on the ocular surface. However, its perioperative utility in cataract surgery has not been formally evaluated.

Eligible participants included consecutive adults (≥18 years) scheduled for phacoemulsification. Key exclusion criteria were a prior diagnosis of ocular surface disease (OSD) or dry eye disease (DED), any history of ocular surgery in either eye, ocular comorbidities, and the current or regular use of topical or instrumental ocular treatments.

Participants were randomized into two groups: the intervention group received LLLT using the Eye-light® device (Espansione Group, Italy), and the control group received sham treatment with an identical, inactive device. Treatments were administered one week before and one week after surgery. The mask delivers light in the 600-1200 nm range through closed eyelids for 15 minutes per session, targeting the periocular region and meibomian glands.

Clinical assessments were performed at baseline (T0), one week postoperatively (T1), one month postoperatively (T2), and six months postoperatively (T3) and included:

* Ocular Surface Disease Index (OSDI)
* Non-invasive tear break-up time (NIBUT)
* Schirmer I test (SIT)
* Corneal fluorescein staining (Oxford grading)
* Tear Osmolarity
* Tear Inflammatory and reparative biomarkers

The primary outcome was the change in OSDI score from baseline to 6 months postoperatively. Secondary outcomes included all objective ocular surface parameters. Safety was evaluated by monitoring treatment-emergent adverse events and assessing patient tolerability of the device.

All surgeries were performed by the same experienced surgeon using standard microincisional phacoemulsification technique. Only eyes without significant intraoperative or postoperative complications were included in the final analysis.

Postoperative therapy was identical for all patients and included a combination of topical dexamethasone and netilmicin for 1 week, followed by tapering dexamethasone alone over 2 additional weeks; topical ketorolac tapered over 3 weeks; and preservative-free artificial tears (cross-linked hyaluronic acid, trehalose, sterilamine in liposomes) administered three times daily for 6 months.

Statistical analysis was performed using SPSS (version 30.0.0.0, SPSS Inc., Chicago, IL, USA).. The normality of data was evaluated using the Shapiro-Wilk test. For normally distributed variables, repeated measures ANOVA followed by Dunnett's post-hoc tests were used. For non-normally distributed data, the Friedman test with Dunn's correction was applied. A p-value < 0.05 was considered statistically significant.

This is the first prospective study to investigate LLLT in the perioperative setting of cataract surgery within consecutive patients. The findings aim to provide evidence for integrating non-pharmacological interventions in ocular surface optimization before and after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult patients (aged ≥18 years).
* Scheduled for routine phacoemulsification cataract surgery.
* Provided written informed consent and agreed to attend all follow-up visits.

Exclusion Criteria:

* Prior diagnosis of ocular surface disease (OSD) or dry eye disease (DED).
* History of ocular surgery in either eye.
* Presence of ocular comorbidities (e.g., glaucoma, uveitis, corneal dystrophies).
* Current or regular use of topical ocular treatments such as lubricants, corticosteroids, or cyclosporine.
* Ongoing or recent instrumental therapies or oral supplements for OSD or DED.
* Use of systemic medications known to be associated with DED (e.g., diuretics, antidepressants, antihistamines, hormone replacement therapy).
* History of autoimmune diseases (e.g., Sjögren's syndrome).
* Regular contact lens wear.
* Any intraoperative or postoperative complications that could interfere with ocular surface evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Baseline to 6 months after cataract surgery
  The Ocular Surface Disease Index (OSDI) is a validated 12-item questionnaire used to assess the severity of dry eye symptoms and their impact on vision-related functioning. The total score ranges from 0 to 100, with higher scores indicating greater symptom severity. Participants will complete the OSDI questionnaire at baseline, 1 week, 1 month, and 6 months postoperatively. The primary outcome is the change in total OSDI score from baseline to 6 months after surgery, comparing the LLLT group to the sham group.

SECONDARY OUTCOMES:
Tear Film Break-Up Time (TBUT) | Baseline to 6 months after cataract surgery
  Tear Film Break-Up Time (TBUT) measures tear film stability by recording the time (in seconds) between a complete blink and the first appearance of a dry spot on the corneal surface after fluorescein dye instillation. Lower TBUT values indicate more severe tear film instability and are commonly used in dry eye diagnosis and monitoring. TBUT will be measured at baseline, 1 week, 1 month, and 6 months following cataract surgery using slit-lamp biomicroscopy and cobalt blue illumination. The change in TBUT from baseline to 6 months postoperatively will be compared between the LLLT and sham groups.
Corneal Fluorescein Staining (CFS) | Baseline to 6 months after cataract surgery
  Corneal fluorescein staining (CFS) is used to assess ocular surface epithelial damage by applying fluorescein dye and evaluating punctate staining patterns under cobalt blue light. The severity is graded using the Oxford grading scale (0-5), with higher scores indicating more extensive corneal damage. CFS will be measured at baseline, 1 week, 1 month, and 6 months after cataract surgery. The secondary outcome is the change in Oxford CFS score from baseline to 6 months, comparing patients receiving low-level light therapy (LLLT) versus sham treatment.
Tear Osmolarity | Baseline to 6 months after cataract surgery
  Tear osmolarity is a core diagnostic biomarker for dry eye disease, reflecting tear film instability and inflammation. Elevated osmolarity values are associated with more severe ocular surface dysfunction. In this study, tear osmolarity will be measured using the TearLab Osmolarity System, a clinically validated point-of-care device that analyzes a 50-nanoliter tear sample from the inferior tear meniscus. Measurements will be taken at baseline, 1 week, 1 month, and 6 months after cataract surgery. The outcome measure is the change in osmolarity values from baseline to 6 months postoperatively, comparing the low-level light therapy (LLLT) and sham groups.
Schirmer I Test | Baseline to 6 months after cataract surgery
  The Schirmer I Test is a standard diagnostic tool used to measure aqueous tear production. Without anesthesia, a sterile paper strip is placed in the lower conjunctival sac for 5 minutes, and the length of the moistened area (in millimeters) indicates tear secretion. Lower values reflect aqueous-deficient dry eye. In this study, the Schirmer I Test will be performed at baseline, 1 week, and 6 months after cataract surgery. The secondary outcome is the change in tear production from baseline to 6 months postoperatively, comparing results between patients treated with low-level light therapy (LLLT) and those receiving sham treatment.
Tear Inflammatory and Reparative Biomarkers | Baseline to 1 month after cataract surgery
  Tear inflammatory and reparative biomarkers are assessed using validated multiplex immunoassays to characterize ocular surface immune and homeostatic status. Platelet-Derived Growth Factor AB (PDGF-AB, normal ≤12.63 pg/mL) and Platelet-Derived Growth Factor CC (PDGF-CC, normal ≤34.96 pg/mL) are evaluated as markers of epithelial repair and tissue remodeling. Vascular Endothelial Growth Factor A (VEGFA, normal ≤4.36 pg/mL) is measured as an indicator of angiogenic activation. Tumor Necrosis Factor alpha (TNF-α, normal ≤3.45 pg/mL) is assessed as a key pro-inflammatory cytokine. Osteopontin (OPN, normal ≤561 pg/mL) and Osteoprotegerin (OPG, normal ≤31.89 pg/mL) are evaluated as modulators of inflammatory balance and tissue integrity. Values above these thresholds are considered suggestive of increased ocular surface inflammation. All biomarkers are measured in both the low-level light therapy (LLLT) group and the sham group at baseline and at 30 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy "Grigore T. Popa" Iași, Iași, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared, including demographic information (age, sex), baseline and follow-up ocular surface parameters (e.g., OSDI scores, tear break-up time, Schirmer I test, corneal staining, tear osmolarity), and treatment adherence data. No personally identifiable information will be disclosed. Data will be made available only upon reasonable request and for research purposes approved by an ethics committee or institutional review board.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Timofte-Zorila MM, Lixi F, Vlas N, Troisi M, Ozkan G, Pavel-Tanasa M, Istrate S, Preda C, Coco G, Namazbayeva A, Giannaccare G, Branisteanu DC. Effect of Low-Level Light Therapy on Ocular Surface Parameters in Patients Undergoing Cataract Surgery: A Prospective Double-Masked Randomized Controlled Clinical Trial. Ophthalmol Ther. 2025 Oct;14(10):2557-2569. doi: 10.1007/s40123-025-01228-6. Epub 2025 Aug 24. PMID 40849606